CLINICAL TRIAL: NCT07343999
Title: A Prospective, Randomized, Multicenter Clinical Trial on the Effect of a Home-Based Multicomponent Exercise Program Combined With Nutritional Supplementation in Patients With Transthyretin Cardiac Amyloidosis
Brief Title: EFICAC-TTR Trial: Exercise and Nutritional Supplementation in Transthyretin Cardiac Amyloidosis
Acronym: EFICAC-TTR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Collaborators: Hospital Universitario de Burgos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFICAC-TTR-UBU-HUBU
Record Dates: First submitted 2025-12-17; First posted 2026-01-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Transthyretin Cardiac Amyloidosis
Keywords: Exercise Training; Nutritional Supplementation; Creatine; Beta-Hydroxy Beta-Methylbutyrate; Older Adults; Functional Capacity; Frailty; Cardiac Amyloidosis; Transthyretin Cardiac Amyloidosis
MeSH Terms: conditions — Frailty; Amyloid Neuropathies, Familial | interventions — microcrystalline cellulose; Creatine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel groups and remain in the assigned group for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The study is open-label. Outcome assessors are blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Other): Participants receive usual medical care for transthyretin cardiac amyloidosis, including routine cardiology follow-up and general lifestyle recommendations, without structured exercise or nutritional supplementation.
  Interventions: Other: Usual Care
- Exercise + Fiber Supplementation (Active Control) (Placebo Comparator): Participants perform a home-based multicomponent exercise program and receive daily supplementation with microcrystalline cellulose, used as a nutritionally inert control supplement.
  Interventions: Behavioral: Home-Based Multicomponent Exercise Program; Dietary Supplement: Fiber Supplementation (Microcrystalline Cellulose)
- Exercise + Creatine and HMB Supplementation (Experimental): Participants perform a home-based multicomponent exercise program and receive daily supplementation with creatine monohydrate (3 g/day) and β-hydroxy-β-methylbutyrate (HMB, 3 g/day).
  Interventions: Behavioral: Home-Based Multicomponent Exercise Program; Dietary Supplement: Creatine and HMB Supplementation

INTERVENTIONS:
Other: Usual Care — Standard clinical management for transthyretin cardiac amyloidosis according to routine cardiology practice.
  Arms: Usual Care
Behavioral: Home-Based Multicomponent Exercise Program — A 12-week home-based multicomponent exercise program adapted from the Vivifrail model, including strength, balance, mobility, and endurance exercises tailored to individual functional capacity.
  Arms: Exercise + Creatine and HMB Supplementation; Exercise + Fiber Supplementation (Active Control)
Dietary Supplement: Fiber Supplementation (Microcrystalline Cellulose) — Daily oral supplementation with microcrystalline cellulose, used as a nutritionally inert control supplement to match supplementation procedures.
  Arms: Exercise + Fiber Supplementation (Active Control)
Dietary Supplement: Creatine and HMB Supplementation — Daily oral supplementation with creatine monohydrate (3 g/day) and β-hydroxy-β-methylbutyrate (HMB, 3 g/day) for 12 weeks.
  Arms: Exercise + Creatine and HMB Supplementation

SUMMARY:
Transthyretin cardiac amyloidosis (TTR-CA) is a heart disease that mainly affects older adults and often leads to reduced physical capacity, muscle weakness, frailty, and a decline in quality of life. While current medical treatments can slow disease progression, they do not fully address functional limitations or muscle deterioration.

The EFICAC-TTR study is a prospective, randomized, multicenter clinical trial designed to evaluate whether a combined non-pharmacological intervention can improve physical function in patients aged 70 years or older with confirmed TTR-CA.

A total of 102 participants will be randomly assigned to one of three groups: (1) usual medical care, (2) a home-based multicomponent exercise program combined with fiber supplementation, or (3) the same exercise program combined with creatine monohydrate and β-hydroxy-β-methylbutyrate (HMB) supplementation. The exercise program is adapted to each participant's functional level and is performed at home.

The main outcomes of the study are changes in walking capacity, measured by the 6-minute walk test, and muscle strength, assessed by handgrip strength after 12 weeks. Secondary outcomes include changes in body composition, frailty, quality of life, and clinical events, while mechanistic biomarkers are assessed as exploratory outcomes.

This study aims to determine whether combining exercise with nutritional supplementation can safely improve functional capacity and overall health in older adults with transthyretin cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years.
* Confirmed diagnosis of transthyretin cardiac amyloidosis (TTR-CA) based on positive bone scintigraphy with diphosphonates (Perugini grade 2 or 3) and absence of monoclonal protein.
* Clinical stability during the 4 weeks prior to enrollment.
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Light-chain (AL) amyloidosis or other non-TTR amyloidosis variants.
* Absolute medical contraindication to moderate-intensity exercise.
* Severe comorbid conditions with an estimated life expectancy <6 months.
* Severe cognitive impairment (Mini-Mental State Examination score <20).
* Concurrent participation in another clinical trial or structured exercise program.
* Known allergy or intolerance to creatine, beta-hydroxy-beta-methylbutyrate (HMB), or microcrystalline cellulose.
* Severe renal impairment requiring dialysis.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Handgrip Strength | Baseline and 12 weeks
  Change in maximal isometric handgrip strength measured in kilograms (kg) using a calibrated handheld dynamometer (best of three attempts for the dominant hand), expressed as the difference between baseline and 12 weeks.
Change in 6-Minute Walk Test Distance | Baseline and 12 weeks
  Change in walking capacity assessed by the 6-minute walk test, measured as the difference in total distance walked (meters) between baseline and 12 weeks.

SECONDARY OUTCOMES:
Change in Fat Mass | Baseline and 12 weeks
  Change in total body fat mass measured in kilograms (kg) using multifrequency bioelectrical impedance analysis, expressed as the difference between baseline and 12 weeks.
Change in Skeletal Muscle Mass | Baseline and 12 weeks
  Change in skeletal muscle mass measured in kilograms (kg) using multifrequency bioelectrical impedance analysis, expressed as the difference between baseline and 12 weeks.
Change in Fat-Free Mass | Baseline and 12 weeks
  Change in fat-free mass measured in kilograms (kg) using multifrequency bioelectrical impedance analysis, expressed as the difference between baseline and 12 weeks.
Change in Phase Angle | Baseline and 12 weeks
  Change in phase angle measured in degrees (°) using multifrequency bioelectrical impedance analysis, expressed as the difference between baseline and 12 weeks.
Change in Frailty Status Assessed by the FRAIL Scale | Baseline and 12 weeks
  Change in frailty status assessed by the FRAIL scale, a 5-item questionnaire with scores ranging from 0 to 5, where higher scores indicate greater frailty, expressed as the difference between baseline and 12 weeks.
All-Cause Mortality | Up to 6 months
  All-cause mortality, defined as death from any cause during the follow-up period.
Change in Short Physical Performance Battery (SPPB) Score | Baseline and 12 weeks
  Change in Short Physical Performance Battery (SPPB) total score, ranging from 0 to 12 points, where higher scores indicate better physical performance, expressed as the difference between baseline and 12 weeks.
Change in Clinical Frailty Scale (CFS) Score | Baseline and 12 weeks
  Change in frailty severity assessed by the Clinical Frailty Scale (CFS), a 9-point ordinal scale ranging from 1 (very fit) to 9 (terminally ill), where higher scores indicate greater frailty.
Change in Barthel Index Score | Baseline and 12 weeks
  Change in functional independence assessed by the Barthel Index, scored from 0 to 100, where higher scores indicate greater independence.
Change in SARC-F Score | Baseline and 12 weeks
  Change in sarcopenia risk assessed by the SARC-F questionnaire, with scores ranging from 0 to 10, where higher scores indicate greater sarcopenia risk.
Change in Minnesota Living With Heart Failure Questionnaire Score | Baseline and 12 weeks
  Change in health-related quality of life assessed by the Minnesota Living With Heart Failure Questionnaire (MLHFQ), with total scores ranging from 0 to 105, where higher scores indicate worse quality of life.
Change in Charlson Comorbidity Index | Baseline and 12 weeks
  Change in comorbidity burden assessed using the Charlson Comorbidity Index, a weighted index that accounts for the number and severity of comorbid conditions, where higher scores indicate greater comorbidity burden.
Incidence of Heart Failure Hospitalizations | Up to 6 months
  Number of hospitalizations due to heart failure occurring during the follow-up period.
Incidence of Non-Heart Failure Hospitalizations | Up to 6 months
  Hospital admissions due to causes other than heart failure during the follow-up period.
Incidence of Emergency Department Visits | Up to 6 months
  Number of emergency department visits during follow-up.
Incidence of Intervention-Related Adverse Events | Up to 6 months
  Number and type of adverse events related to exercise and/or supplementation, classified according to severity and relatedness, collected throughout the follow-up period.
Rate of Supplement Discontinuation | Up to 6 months
  Proportion of participants who discontinue study supplements.
Exercise Program Adherence | Up to 12 weeks
  Proportion (%) of prescribed exercise sessions completed, with adequate adherence defined as completion of at least 80% of prescribed sessions.
Supplement Adherence | Up to 12 weeks
  Proportion (%) of planned supplement doses consumed, with optimal compliance defined as 90-110%.

OTHER OUTCOMES:
Change in Growth Differentiation Factor 15 (GDF-15) | Baseline and 12 weeks
  Change in serum GDF-15 concentration (pg/mL) measured by immunoassay.
Change in Soluble ST2 | Baseline and 12 weeks
  Change in serum soluble ST2 concentration (ng/mL) measured by immunoassay.
Change in Interleukin-6 (IL-6) | Baseline and 12 weeks
  Change in serum interleukin-6 (IL-6) concentration (pg/mL) measured by immunoassay.
Change in C-Reactive Protein (CRP) | Baseline and 12 weeks
  Change in serum C-reactive protein (CRP) concentration (mg/L) measured by immunoassay.
Change in circulating miR-21 expression | Baseline and 12 weeks
  Change in circulating miR-21 expression measured by quantitative PCR, expressed as relative expression (ΔΔCt).
Change in circulating miR-29 expression | Baseline and 12 weeks
  Change in circulating miR-29 expression measured by quantitative PCR, expressed as relative expression (ΔΔCt).
Change in circulating miR-34a expression | Baseline and 12 weeks
  Change in circulating miR-34a expression measured by quantitative PCR, expressed as relative expression (ΔΔCt).
Change in circulating miR-155 expression | Baseline and 12 weeks
  Change in circulating miR-155 expression measured by quantitative PCR, expressed as relative expression (ΔΔCt).
Change in PBMC Macrophage Polarization (M1/M2) by Flow Cytometry | Baseline and 12 weeks
  Change in macrophage polarization profile assessed by flow cytometry immunophenotyping of PBMC-derived macrophages, expressed as M1/M2 ratio.
Change in Pro-inflammatory (M1) Gene Expression Markers | Baseline and 12 weeks
  Change in gene expression of predefined pro-inflammatory (M1) markers in PBMC-derived macrophages, measured by quantitative PCR and expressed as relative expression (ΔΔCt).
Change in Anti-inflammatory (M2) Gene Expression Markers | Baseline and 12 weeks
  Change in gene expression of predefined anti-inflammatory (M2) markers in PBMC-derived macrophages, measured by quantitative PCR and expressed as relative expression (ΔΔCt).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Mielgo-Ayuso, PhD, Principal Investigator — Universidad de Burgos; José A Pérez Rivera, PhD, MD, Study Chair — Hospital Universitario de Burgos

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication and ending 5 years after publication.
Access Criteria: Access to de-identified individual participant data will be granted upon reasonable request to the principal investigator. Requests must include a methodologically sound research proposal and will be evaluated for scientific merit and feasibility. Data sharing will require the execution of a data sharing agreement and will comply with applicable data protection and privacy regulations.

REFERENCES:
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Result] Ramos-Hernandez R, Miguel-Ortega A, Martinez-Ferran M, Fernandez-Lazaro D, Busto N, Mielgo-Ayuso J. Combined creatine and HMB co-supplementation improves functional strength independent of muscle mass in physically active older adults: a randomized crossover trial. Geroscience. 2025 Oct 10. doi: 10.1007/s11357-025-01889-y. Online ahead of print. PMID 41073834
- [Result] de Souto Barreto P, Rolland Y, Vellas B, Maltais M. Association of Long-term Exercise Training With Risk of Falls, Fractures, Hospitalizations, and Mortality in Older Adults: A Systematic Review and Meta-analysis. JAMA Intern Med. 2019 Mar 1;179(3):394-405. doi: 10.1001/jamainternmed.2018.5406. PMID 30592475
- [Result] Garcia-Pavia P, Rapezzi C, Adler Y, Arad M, Basso C, Brucato A, Burazor I, Caforio ALP, Damy T, Eriksson U, Fontana M, Gillmore JD, Gonzalez-Lopez E, Grogan M, Heymans S, Imazio M, Kindermann I, Kristen AV, Maurer MS, Merlini G, Pantazis A, Pankuweit S, Rigopoulos AG, Linhart A. Diagnosis and treatment of cardiac amyloidosis: a position statement of the ESC Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2021 Apr 21;42(16):1554-1568. doi: 10.1093/eurheartj/ehab072. PMID 33825853
- [Result] Ruberg FL, Grogan M, Hanna M, Kelly JW, Maurer MS. Transthyretin Amyloid Cardiomyopathy: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Jun 11;73(22):2872-2891. doi: 10.1016/j.jacc.2019.04.003. PMID 31171094